CLINICAL TRIAL: NCT02740595
Title: The Effects of Electronic Cigarettes on Endothelial Function and Oxidative Stress
Brief Title: E-cigarettes and Blood Vessel Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Holly R Middlekauff, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14-000743
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Nicotine Dependence
Keywords: nicotine; endothelial function; oxidative stress
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nicotine (Experimental): Use an e-cig filled with liquid with nicotine
  Interventions: Other: one time exposure to e-cig with nicotine
- no nicotine (Experimental): Use an e-cig filled with liquid without nicotine
  Interventions: Other: one time exposure to e-cig without nicotine
- sham comparator (Sham Comparator): Use an empty e-cigarette (sham control)
  Interventions: Other: one time exposure to empty e-cig

INTERVENTIONS:
Other: one time exposure to e-cig with nicotine — one time exposure to e-cig vapor with nicotine
  Arms: Nicotine
Other: one time exposure to e-cig without nicotine — one time exposure to e-cig without nicotine
  Arms: no nicotine
Other: one time exposure to empty e-cig — one time exposure to empty e-cig (sham control
  Other Names: sham control
  Arms: sham comparator

SUMMARY:
Randomized controlled trial of electronic cigarettes with nicotine, without nicotine, and sham control, on endothelial function and markers of oxidative stress.

DETAILED DESCRIPTION:
Participants will use an electronic cigarette on 3 occasions: 1) with nicotine, 2) without nicotine, 3) sham control, and undergo a measure of endothelial function called brachial artery flow mediated dilatation (FMD). Additionally, oxidative stress will be measured pre and post exposure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Cardiac disease
* Respiratory disease
* Diabetes mellitus

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2015-08; Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilatation (FMD) | 10 minutes after exposure
  FMD is a measure of endothelial function
Paraoxonse | less than 1 hour after exposure
  plasma oxidative stress

CONTACTS AND LOCATIONS:
Locations (1):
- UCaliforniaLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No